CLINICAL TRIAL: NCT00769106
Title: A Randomized Controlled Study of Cytokine-induced Killer Cell (CIK) Treatment in Patients With Hepatocellular Carcinoma Who Underwent Radical Resection.
Brief Title: Study of Cytokine-induced Killer Cell (CIK) Treatment in Patients After Resection of Liver Cancer
Acronym: HCC-CIK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, LI Sheng-ping, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-senU 5010
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2015-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; recurrent; cytokine-induced killer cell
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (control group) (No Intervention): regular treatment and follow up
- A (CIK group) (Experimental): cytokine-induced killer cell treatment plus regular treatment and follow up
  Interventions: Biological: cytokine-induced killer cell (CIK) treatment

INTERVENTIONS:
Biological: cytokine-induced killer cell (CIK) treatment — cytokine-induced killer cell treatment every two weeks, for 4 cycles
  Other Names: CIK
  Arms: A (CIK group)

SUMMARY:
Study hypothesis:

The recurrence rate of HCC patients after radical resection is about 60-70%. This study is based on the hypothesis that CIK treatment could decrease the recurrence rate by 15% to 20%.

Abstract:

This is a randomized controlled study. About 200 patients with hepatocellular carcinoma who underwent radical resection will be included. The patients will be randomized to group A (receive CIK treatment) or group B (just regularly follow up) without any anti-cancer treatment after resection of HCC, and the randomize ratio will be 1:1.

Study treatment:

Patients in group A will receive 4 cycles of CIK treatments within 3 months after their liver resection. Patients in group B will have no anti-cancer therapy. Anti-virus and other supportive therapies are available in both groups.

ELIGIBILITY:
Inclusion Criteria

* Male or female patients > 18 years of age.
* Without any prior anti-cancer therapy.
* Patients who have a life expectancy of at least 12 weeks.
* Patients already had radical resection of HCC.
* Definition of radical resection in this study:
* All tumors were moved out, with a clean resection margin.
* Number of tumors <= 3.
* Without tumor invasion of the main trunk and first branch of the portal vein, or hepatic duct, or hepatic vein.
* No hepatic hilum lymphnode metastasis.
* No distance metastasis.
* Hepatocellular carcinoma with histological diagnose.
* No major post-operative complication.
* Patients who have an ECOG PS of 0, or 1.
* Cirrhotic status of Child-Pugh class A only.
* The following laboratory parameters:

  * Platelet count >= 70 x 109/L
  * Hemoglobin >= 8.5 g/dL
  * Albumin >= 3.5 g/dL
  * Total bilirubin <= 25umol/L
  * Alanine transaminase (ALT) and AST <= 2.5 x upper limit of normal
  * Serum creatinine <= 1.5 x the upper limit of normal
  * Prothrombin time (PT) <= 3 seconds above control.
  * Patients who give written informed consent.

Exclusion Criteria

* Previous or concurrent cancer that is distinct in primary site or histology from HCC.
* History of cardiac disease.
* Active clinically serious infections (> grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* History of organ allograft.
* Known or suspected allergy to the investigational agent or any agent given in association with this trial.
* Pregnant or breast-feeding patients.
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study.

Excluded therapies and medications, previous and concomitant:

* Prior use of any anti-cancer treatment for HCC, eg. chemotherapy, radiotherapy.
* Antiviral treatment is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to recurrence (TTR) | month

SECONDARY OUTCOMES:
Overall survival (OS) | month
Progression Free Survival (PFS) | month
Laboratory findings | every 3 months
AEs and SAEs | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Jin-qing Li, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China